CLINICAL TRIAL: NCT06128655
Title: Developing and Testing a Nurse-Led Technology-Enhanced Family Engagement Program (NURSE-TECH-Family) Among Critically Ill Patients in ICU: A Randomized Controlled Trial
Brief Title: Developing and Testing a Nurse-Led Technology-Enhanced Family Engagement Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Brigitte S. Cypress, EdD, RN, CCRN, ASSOCIATE PROFESSOR, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2023000214; Registration No. IORG0000357 (Other: Rutgers University)
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP: survey and Standard Care (SC) or no NURSE-TECH-Family during PFCC-IR participation (No Intervention): 15 family members
- EXPERIMENTAL GROUP: participation in NURSE-TECH-Family during PFCC-IR (Experimental): 15 family members
  Interventions: Other: Participation in PFCC-IR

INTERVENTIONS:
Other: Participation in PFCC-IR — PFCC-IR with the critical care team is standard practice in ICU but it doesn't usually include family members. The intervention for this study is interdisciplinary patient care rounds that include one family member of the patient.
  Arms: EXPERIMENTAL GROUP: participation in NURSE-TECH-Family during PFCC-IR

SUMMARY:
Family engagement in care for ICU patients is essential to ensure patient-centered clinical outcomes such as reducing ICU length of stay (LOS) by about a day, and hospital LOS from 3.78 days to 2.29 days. It also lowers patient's stress and anxiety, improves orientation, and detection, lowers the prevalence and duration of delirium; enhances patients' and families' satisfaction and experience with care and helps with patients' recovery. This practice has not been universally implemented due to issues with lack of transportation for family members to the hospital, time conflict with work, and clinicians' fear of engaging family. Family-centered care in the ICU remains an inconsistent practice and an understudied area of nursing science. Family-centered care in the ICU remains an inconsistent practice and an understudied area of nursing science. The purpose of this proposed study is to determine the feasibility of conducting a randomized controlled trial (RCT) to implement and test the impact of a Nurse-Led-Technology-EnhanCed Family Engagement Program (Nurse-TECH-Family) on the primary outcome of ICU LOS, and secondary outcome of reducing stress and improving quality of life and well-being among critically ill patients' families. We propose a pilot two-group RCT to examine the feasibility and preliminary effects of NURSE-TECH-Family program on 30 family members in the ICU. This study will be conducted at the Cooper University Health Care Medical Intensive Care Unit. Prior to conducting the RCT, we will involve a focus group of eight healthcare providers to understand healthcare providers' perceptions of the intervention and the project. The specific aims of this RCT are to (1) Assess the feasibility and acceptability of NURSE-TECH-Family program and obtain data on family stress, mental and physical health symptoms, and quality of life of family members. (2) Provide preliminary data for estimation of the effects of NURSE-TECH-Family program on family stress, mental and physical health symptoms, and quality of life post-program compared to a control group who will receive the current standard care. (3) Explore the effects of NURSE-TECH-Family on LOS and satisfaction based on Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) scores at post-program compared to a control group who will receive the current standard care.

DETAILED DESCRIPTION:
Purpose/Specific Aims The overall goal of our research is to test the impact of Nurse-TECH-Family program during patient-and-family-centered interdisciplinary rounds (PFCC-IR) in the ICU. Our central hypothesis is that the use of nurse liaisons who utilize telehealth technology to target the barriers to family-engaged critical care (e.g., transportation, time constraints, work-obligations) would lead to less stress and mental and physical health symptoms, and improved quality of life among family members of patients in critical care.

Research Design We propose a pilot two-group RCT to examine the feasibility and preliminary effects of the NURSE-TECH-Family program on 30 family members in the ICU. This study will be conducted at the Cooper University Health Care Intensive Care Unit. Prior to conducting the RCT, we will involve a focus group of eight healthcare providers to understand healthcare providers' perception of the intervention and the project

A. Objectives Aim 1: Assess the feasibility and acceptability of the Nurse-TECH-Family program and obtain data on family stress, mental and physical health symptoms, and the quality of life of family members. Feasibility will be assessed using study accrual, protocol adherence, and retention.

Aim 2: Provide preliminary data for estimating the effects of the Nurse-TECH-Family program on family stress, mental and physical health symptoms, and quality of life at post-program compared to the control group who will receive the current standard care (SC).

Aim 3: Explore the effects of Nurse-TECH-Family on LOS and satisfaction based on Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) scores at post-program compared to a control group who will receive the current standard care.

B. Hypotheses / Research Question(s) H1: Feasibility will be determined by >80% adherence to the protocol, and <20% attrition. Acceptability will be demonstrated by 80% of participants reporting intervention satisfaction.

H2: Between-group effect sizes will be used to evaluate intervention efficacy on measures of stress, mental and physical health symptoms, and quality of life.

H3: Between-group effect sizes will be used to evaluate patterns suggesting intervention efficacy on LOS and satisfaction based on HCAHPS scores at post-program compared to a control group who will receive the current standard care. This study is not designed to make conclusions about efficacy without further study.

Study Variables A. Independent Variables, Interventions, or Predictor Variables Intervention: participation in Nurse-TECH-Family during PFCC-IR participation; Control: Standard Care (SC) or no Nurse-TECH-Family during PFCC-IR participation

B. Dependent Variables or Outcome Measures Outcome 1: number of days for ICU stay; Outcome 2/Secondary Outcomes: physical symptoms in gastrointestinal, respiratory, neurological, cognitive, sleep, swallowing/voice body system; Outcome 3: mental symptoms (depression, anxiety, and stress)

Study Population The eight (8) healthcare providers will include nurses and physicians between 25-80 years old working in the CCU who are willing to participate in focus group sessions.

Family members:

Inclusion criteria: (1) men and women 18-80 years old who are willing to participate in Nurse-TECH Family.

Exclusion criteria: (1) men and women who are under 18 or over 80 years old who are not willing to participate in Nurse-TECH Family.

Research Procedures This feasibility study will help us provide preliminary data for a bigger study, assess the viability of the research plan, and evaluate the adequacy and practicality of the logistics required for delivering the planned intervention and the application of research methods, rather than looking for significance.

Following consent, 30 participants will be randomly assigned in equal allocation to one of two conditions: 1) participation in Nurse-TECH-Family intervention or 2) standard care (SC). The data manager on this study who is not involved with recruitment will randomly draw a number of 1 or 2 to be given the participant's study number (not name) to randomize the participant. Our research evaluator will not be involved in recruitment or have any contact with participants; they will be blinded to participant randomization and conduct all study procedures where blinding is indicated.

RCT Randomization: Following consent, 30 participants will be randomly assigned in equal allocation to one of two conditions: 1) participation in Nurse-TECH-Family intervention or 2) standard care (SC). The data programmer in this study who is not involved with recruitment will randomly draw a number of 1 or 2 to be given the participant's study number (not name) to randomize the participant. Our research evaluator will not be involved in recruitment or have any contact with participants; they will be blinded to participant randomization and conduct all study procedures where blinding is indicated).

Treatment Conditions: Patient-and-family-centered care interdisciplinary rounds (PFCC-IR) are walking rounds - a key strategy for ensuring that the entire team is involved in the care coordination process and that these interventions take place in a timely manner. It is led by the CCU Attending and consists of other members of the medical team assigned to the CCU such as interns, medical residents, fellows, nurses, nurse managers, and other health care professionals such as respiratory therapists and dietitians. A family member and/or significant other will be present to attend this round if they are present in the CCU. The focus of PFCC-IR is to discuss the patient's present condition and plan of care, expected outcomes of care including prognosis, barriers, and challenges to care, transitions in care, and transfer or discharge plan from CCU.

Participants in the Nurse-TECH Family group are expected to participate daily in PFCC-IR when present in CCU. For family members who are not in the CCU in person, the nurse (PIs) will call or virtually via Webex or Microsoft Teams with them daily after the PFCC-IR. The participants in the control group will get SC.

Data Points Participants will have two to complete study assessment measures: baseline, demographic, and social variables (day 1 when in the study) and post-Nurse-TECH Family (when patients leave the CCU). The research evaluator who will be blinded to the group allocation will collect data.

Feasibility will be assessed by examining study accrual, protocol adherence, and retention.

During Study Data:

Baseline (day 1 when in the study) and post-intervention data (when patients leave the CCU):

Demographic, Social, and Medical Variables will be collected via family member's self-report including age, gender, education level, occupational status, socioeconomic determinants of health, and caregiver.

Physical symptoms. The Symptom Experience Index assesses 20 symptoms that indicate the physiological changes in gastrointestinal, respiratory, neurological, cognitive, sleep, swallowing/voice body system (Cronbach's alpha of 0.85 -0.86).

Mental health symptoms. The 2-item Patient Health Questionnaire screen tool with a sensitivity=100% (specificity=77%, AUC=0.88) will be used to assess depression; The Generalized Anxiety Disorder 2-item screen tool with a sensitivity=86% (specificity=83%, Positive likelihood ratio=5.0) will be used to assess anxiety (Cronbach's greater than .70).

Quality of life (QOL). The Short-Form Health Survey (SF-36), a valid and reliable tool, will be used to assess QOL (24). The SF-36 included 8 subscales: (1) physical functioning; (2) role physical, i.e. role limitations because of physical problems; (3) bodily pain; (4) general health; (5) social functioning; (6) role emotional, i.e. role limitations because of emotional problems; (7) vitality (energy/fatigue); (8) mental health, i.e. psychological distress and psychological well-being.

Socioeconomic determinants. Items to screen for social needs and financial strains in The Accountable Health Communities (AHC) model will be used to assess socioeconomic determinants. Demographic and Health Characteristics. Demographic and health characteristics will be assessed using The Accountable Health Communities (AHC) model to include age, gender, race/ethnicity, employment, education, number of chronic conditions, physical activity, substance use, disability, and income.

Study Duration The study duration for each participant is during the CCU stay (a few days to about a week, and 40-45 minutes for assessment on day 1 and the day the patient leaves the CCU). The study duration for the healthcare providers in the focus group will be 2-3 hours.

Sample Size Justification This is a pilot two-group randomized controlled trial to examine the feasibility and preliminary effects of the Nurse-TECH Family program on 30 family members of critically ill patients in the CCU. We are aiming to consecutively recruit a sample size of 30, 15 in each arm. Assuming an effect size of 30 (15 per group) is needed. Furthermore, with a sample of 24 patients total, we will generate sufficient data to approximate the first and second moments of the data distributions for the second and third outcome measures to plan a well-powered future study of a similar population.

Location: Data collection will occur in Cooper University Health Care (Cooper) CCU.

Timing and Frequency:

Family members: Demographics and baseline data will be collected at Cooper University Health Care (Cooper) on day 1 while the patient is in CCU. Participants will be asked to complete the second assessment when the patient leaves the CCU.

Study Instruments:

Length of stay and satisfaction will be assessed based on Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) scores at post-program.

Physical symptoms. The Symptom Experience Index assesses 20 symptoms that indicate the physiological changes Mental health symptoms. The 2-item Patient Health Questionnaire screen tool with a sensitivity=100% (specificity=77%, AUC=0.88) will be used to assess depression; The Generalized Anxiety Disorder 2-item screen tool with a sensitivity=86% (specificity=83%, Positive likelihood ratio=5.0) will be used to assess anxiety. The 1-item Perceived Stress Scale will be used to assess perceived stress (Cronbach's greater than .70).

Quality of life (QOL). The Short- Form Health Survey (SF-36), a valid and reliable tool, will be used to assess QOL.

Socioeconomic determinants. Items to screen for social needs and financial strains in The Accountable Health Communities (AHC) model will be used to assess socioeconomic determinants.

Data Analysis Aim 1 Analysis. For Aims 1, 2, and 3, Feasibility will be assessed by examining accrual, adherence, and attrition. Accrual will be indicated by meeting the recruitment goal of 30 participants in 12 months. Adherence will be indicated by ensuring stable unit treatment values between the group randomized to the NURSE-TECH Family intervention vs. the control (i.e. no crossover/contamination between groups). Attrition will be indicated by 80% of consented participants completing the study protocol (i.e., remain enrolled and completing questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* men between 18-80 years old who are willing to participate in NURSE-TECH Family
* women between 18-80 years old who are willing to participate in NURSE-TECH Family

Exclusion Criteria:

* men younger than 18 or older than 80 who are not willing to participate in NURSE-TECH Family and are non-English speaking.
* women younger than 18 or older than 80 who are not willing to participate in NURSE-TECH Family and are non-English speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Assessing length of stay (LOS) after Inclusion in PFCC-IR | Post-intervention data (when patients leave the ICU). The data about the number of days in ICU will be assessed upon survey of family members once the patient is discharged from the ICU up to 4 weeks.
  length of stay
Assessing physical symptoms in gastrointestinal, respiratory, neurological, cognitive, sleep, swallowing/voice body system | Baseline (day 1 when in the study) and post-intervention data (when patients leave the ICU) up to 4 weeks.
  Numbers of Health Symptoms. The Symptom Experience Index will measure the number of physical symptoms. This instrument assesses 20 symptoms that indicate the physiological changes in gastrointestinal, respiratory, neurological, cognitive, sleep, swallowing/voice body systems. This reliable and valid tool can differentiate healthy individuals from cancer, medical-surgical, and obstetric patients (Cronbach's alpha = 0.85 -0.86). The instrument uses a Likert scale between 0-5 (never, seldom, frequently, usually, always).
Assessing mental health symptoms: depression | Family members will be surveyed about how often they have been bothered by the symptoms in the last 2 weeks. A post-intervention survey will be administered once the patient leaves the ICU up to 4 weeks
  The 2-item Patient Health Questionnaire (PHQ-2) screen tool with a reported sensitivity=100% (specificity=77%, AUC=0.88) will be used to assess depression. The instrument uses a Likert scale between 0-3 (not at all, several days, more than half the days, nearly every day).
Assessing mental health symptoms: anxiety | Family members will be surveyed about how often they have been bothered by the symptoms in the last 2 weeks. A post-intervention survey will be administered once the patient leaves the ICU up to 4 weeks
  Anxiety: The generalized Anxiety Disorder 2-item (GAD-2) screen tool with a reported sensitivity=86% (specificity=83%, Positive likelihood ratio=5.0) will be used to assess anxiety. The instrument uses a Likert scale between 0-3 (not at all, several days, more than half the days, nearly every day).

CONTACTS AND LOCATIONS:
Overall Officials: BRIGITTE S CYPRESS, Principal Investigator — RUTGERS SCHOOL OF NURSING CAMDEN
Locations (1):
- Cooper University Health Care, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results that will be reported in future articles based on this study will be available after deidentification (texts, tables, figures, and appendices)
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact: brigitte.cypress@rutgers.edu

REFERENCES:
- [Background] Elcokany, N. & Abdel Wareth, M. (2019). Perception of intensive care unit nurses toward family engagement in patients' care. International Journal of Novel Research in Nursing, 6(2), 1099-1110.
- [Background] Goldfarb MJ, Bechtel C, Capers Q 4th, de Velasco A, Dodson JA, Jackson JL, Kitko L, Pina IL, Rayner-Hartley E, Wenger NK, Gulati M; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Lifelong Congenital Heart Disease and Heart Health in the Young; Council on Cardiovascular Radiology and Intervention; Council on Hypertension; Council on the Kidney in Cardiovascular Disease; and Council on Lifestyle and Cardiometabolic Health. Engaging Families in Adult Cardiovascular Care: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2022 May 17;11(10):e025859. doi: 10.1161/JAHA.122.025859. Epub 2022 Apr 21. PMID 35446109
- [Background] Lee HW, Park Y, Jang EJ, Lee YJ. Intensive care unit length of stay is reduced by protocolized family support intervention: a systematic review and meta-analysis. Intensive Care Med. 2019 Aug;45(8):1072-1081. doi: 10.1007/s00134-019-05681-3. Epub 2019 Jul 3. PMID 31270579
- [Background] Rosa RG, Tonietto TF, da Silva DB, Gutierres FA, Ascoli AM, Madeira LC, Rutzen W, Falavigna M, Robinson CC, Salluh JI, Cavalcanti AB, Azevedo LC, Cremonese RV, Haack TR, Eugenio CS, Dornelles A, Bessel M, Teles JMM, Skrobik Y, Teixeira C; ICU Visits Study Group Investigators. Effectiveness and Safety of an Extended ICU Visitation Model for Delirium Prevention: A Before and After Study. Crit Care Med. 2017 Oct;45(10):1660-1667. doi: 10.1097/CCM.0000000000002588. PMID 28671901
- [Background] Jaberi AA, Zamani F, Nadimi AE, Bonabi TN. Effect of family presence during teaching rounds on patient's anxiety and satisfaction in cardiac intensive care unit: A double-blind randomized controlled trial. J Educ Health Promot. 2020 Jan 30;9:22. doi: 10.4103/jehp.jehp_417_19. eCollection 2020. PMID 32154317
- [Background] Heydari A, Sharifi M, Moghaddam AB. Family participation in the care of older adult patients admitted to the intensive care unit: A scoping review. Geriatr Nurs. 2020 Jul-Aug;41(4):474-484. doi: 10.1016/j.gerinurse.2020.01.020. Epub 2020 Feb 12. PMID 32059826
- [Background] Kleinpell R, Zimmerman J, Vermoch KL, Harmon LA, Vondracek H, Hamilton R, Hanson B, Hwang DY. Promoting Family Engagement in the ICU: Experience From a National Collaborative of 63 ICUs. Crit Care Med. 2019 Dec;47(12):1692-1698. doi: 10.1097/CCM.0000000000004009. PMID 31567354
- [Background] Pun BT, Badenes R, Heras La Calle G, Orun OM, Chen W, Raman R, Simpson BK, Wilson-Linville S, Hinojal Olmedillo B, Vallejo de la Cueva A, van der Jagt M, Navarro Casado R, Leal Sanz P, Orhun G, Ferrer Gomez C, Nunez Vazquez K, Pineiro Otero P, Taccone FS, Gallego Curto E, Caricato A, Woien H, Lacave G, O'Neal HR Jr, Peterson SJ, Brummel NE, Girard TD, Ely EW, Pandharipande PP; COVID-19 Intensive Care International Study Group. Prevalence and risk factors for delirium in critically ill patients with COVID-19 (COVID-D): a multicentre cohort study. Lancet Respir Med. 2021 Mar;9(3):239-250. doi: 10.1016/S2213-2600(20)30552-X. Epub 2021 Jan 8. PMID 33428871
- [Background] Kotfis K, Williams Roberson S, Wilson JE, Dabrowski W, Pun BT, Ely EW. COVID-19: ICU delirium management during SARS-CoV-2 pandemic. Crit Care. 2020 Apr 28;24(1):176. doi: 10.1186/s13054-020-02882-x. PMID 32345343
- [Background] Roze des Ordons AL, Au S, Blades K, Stelfox HT. Family participation in ICU rounds-Working toward improvement. J Eval Clin Pract. 2020 Dec;26(6):1620-1628. doi: 10.1111/jep.13345. Epub 2020 Jan 9. PMID 31916653
- [Background] Hetland B, McAndrew N, Perazzo J, Hickman R. A qualitative study of factors that influence active family involvement with patient care in the ICU: Survey of critical care nurses. Intensive Crit Care Nurs. 2018 Feb;44:67-75. doi: 10.1016/j.iccn.2017.08.008. Epub 2017 Nov 21. PMID 29169879
- [Background] Hwang DY, Zhang Q, Andrews A, LaRose K, Gonzalez M, Harmon L, Vermoch K. The Initial Impact of the Coronavirus Disease 2019 Pandemic on ICU Family Engagement: Lessons Learned From a Collaborative of 27 ICUs. Crit Care Explor. 2021 Apr 2;3(4):e0401. doi: 10.1097/CCE.0000000000000401. eCollection 2021 Apr. PMID 33834173
- [Background] Hart JL, Taylor SP. Family Presence for Critically Ill Patients During a Pandemic. Chest. 2021 Aug;160(2):549-557. doi: 10.1016/j.chest.2021.05.003. Epub 2021 May 8. PMID 33971149
- [Background] Hamilton R, Kleinpell R, Lipman J, Davidson JE. International facilitators and barriers to family engagement in the ICU: Results of a qualitative analysis. J Crit Care. 2020 Aug;58:72-77. doi: 10.1016/j.jcrc.2020.04.011. Epub 2020 Apr 22. PMID 32361221
- [Background] Taylor SP, Short RT 3rd, Asher AM, Taylor B, Beidas RS. A rapid pre-implementation evaluation to inform a family engagement navigator program during COVID-19. Implement Sci Commun. 2020 Dec 9;1(1):110. doi: 10.1186/s43058-020-00098-2. PMID 33298192
- [Background] Stücker, O.; Pons-Himbert, C.; Laemmel, E. Towards a better understanding of lymph circulation. Phlebolymphology 2008, 15, 31-36.
- [Background] The University of Texas MD Anderson Cancer Center. November 2019: Exercise and the Lymphatic System. Available online: https://www.mdanderson.org/publications/focused-on-health/exercise-and-the-lymphatic-system.h20-1592991.html (accessed on 10 April 2022).
- [Background] Fu MR, McTernan ML, Qiu JM, Ko E, Yazicioglu S, Axelrod D, Guth A, Fan Z, Sang A, Miaskowski C, Wang Y. The Effects of Kinect-Enhanced Lymphatic Exercise Intervention on Lymphatic Pain, Swelling, and Lymph Fluid Level. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211026757. doi: 10.1177/15347354211026757. PMID 34160294
- [Background] Fu MR, Axelrod D, Guth AA, Scagliola J, Rampertaap K, El-Shammaa N, Qiu JM, McTernan ML, Frye L, Park CS, Yu G, Tilley C, Wang Y. A Web- and Mobile-Based Intervention for Women Treated for Breast Cancer to Manage Chronic Pain and Symptoms Related to Lymphedema: Results of a Randomized Clinical Trial. JMIR Cancer. 2022 Jan 17;8(1):e29485. doi: 10.2196/29485. PMID 35037883
- [Background] Liu F, Li F, Fu MR, Zhao Q, Wang Y, Pang D, Yang P, Jin S, Lu Q. Self-management Strategies for Risk Reduction of Subclinical and Mild Stage of Breast Cancer-Related Lymphedema: A Longitudinal, Quasi-experimental Study. Cancer Nurs. 2021 Nov-Dec 01;44(6):E493-E502. doi: 10.1097/NCC.0000000000000919. PMID 34694088
- [Background] Fu MR, Axelrod D, Guth AA, Cartwright F, Qiu Z, Goldberg JD, Kim J, Scagliola J, Kleinman R, Haber J. Proactive approach to lymphedema risk reduction: a prospective study. Ann Surg Oncol. 2014 Oct;21(11):3481-9. doi: 10.1245/s10434-014-3761-z. Epub 2014 May 9. PMID 24809302
- [Background] Fu MR, Axelrod D, Guth AA, Rampertaap K, El-Shammaa N, Hiotis K, Scagliola J, Yu G, Wang Y. mHealth self-care interventions: managing symptoms following breast cancer treatment. Mhealth. 2016 Jul;2:28. doi: 10.21037/mhealth.2016.07.03. Epub 2016 Jul 22. PMID 27493951
- [Background] Fu MR, Axelrod D, Guth AA, Wang Y, Scagliola J, Hiotis K, Rampertaap K, El-Shammaa N. Usability and feasibility of health IT interventions to enhance Self-Care for Lymphedema Symptom Management in breast cancer survivors. Internet Interv. 2016 Sep;5:56-64. doi: 10.1016/j.invent.2016.08.001. Epub 2016 Aug 4. PMID 28255542
- [Background] Chiang AT, Chen Q, Wang Y, Fu MR. Kinect-Based In-Home Exercise System for Lymphatic Health and Lymphedema Intervention. IEEE J Transl Eng Health Med. 2018 Oct 12;6:4100313. doi: 10.1109/JTEHM.2018.2859992. eCollection 2018. PMID 30456001
- [Background] Chiang AT, Chen Q, Wang Y, Fu MR. Motion Sequence Alignment for A Kinect-Based In-Home Exercise System for Lymphatic Health and Lymphedema Intervention. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:2072-2075. doi: 10.1109/EMBC.2018.8512635. PMID 30440810
- [Background] Chiang AT, Chen Q, Li S, Wang Y, Fu M. Denoising of Joint Tracking Data by Kinect Sensors Using Clustered Gaussian Process Regression. MMHealth17 (2017). 2017 Oct;2017:19-25. doi: 10.1145/3132635.3132642. PMID 30882097
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Miller WL. Fluid Volume Overload and Congestion in Heart Failure: Time to Reconsider Pathophysiology and How Volume Is Assessed. Circ Heart Fail. 2016 Aug;9(8):e002922. doi: 10.1161/CIRCHEARTFAILURE.115.002922. PMID 27436837
- [Background] Lee YW, Jeng YJ, Huang LH. Development and testing of a scale to assess fluid overload symptoms. Appl Nurs Res. 2015 May;28(2):206-9. doi: 10.1016/j.apnr.2014.10.001. Epub 2014 Oct 13. PMID 25457273
- [Background] Pellicori P, Kaur K, Clark AL. Fluid Management in Patients with Chronic Heart Failure. Card Fail Rev. 2015 Oct;1(2):90-95. doi: 10.15420/cfr.2015.1.2.90. PMID 28785439
- [Background] Cooper LB, Lippmann SJ, DiBello JR, Gorsh B, Curtis LH, Sikirica V, Hernandez AF, Sprecher DL, Laskey WK, Saini R, Fonarow GC, Hammill BG. The Burden of Congestion in Patients Hospitalized With Acute Decompensated Heart Failure. Am J Cardiol. 2019 Aug 15;124(4):545-553. doi: 10.1016/j.amjcard.2019.05.030. Epub 2019 May 25. PMID 31208702
- [Background] Parrinello G, Greene SJ, Torres D, Alderman M, Bonventre JV, Di Pasquale P, Gargani L, Nohria A, Fonarow GC, Vaduganathan M, Butler J, Paterna S, Stevenson LW, Gheorghiade M. Water and sodium in heart failure: a spotlight on congestion. Heart Fail Rev. 2015 Jan;20(1):13-24. doi: 10.1007/s10741-014-9438-7. PMID 24942806
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476

DOCUMENTS (1):
  • Informed Consent Form (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT06128655/ICF_000.pdf